CLINICAL TRIAL: NCT04341961
Title: Observational Pilot Study on Pomegranate Metabolism in Breastfeeding Women and Their Infants
Brief Title: Effect of Pomegranate Juice Consumption on the Health of Mothers and Infants During Breastfeeding
Acronym: PomInfant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-001683
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Breastfeeding
Keywords: microbiome; pomegranate; breastmilk
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pom Juice (Experimental): The study participants will all be asked to drink pomegranate juice for 2 weeks, and 4 weeks of continued usual diet and avoid pomegranate juice (other than what is given to you), berries (strawberries, blackberries, raspberries (red, black, yellow), cranberries), walnuts, pecans, hazelnuts, pecans, chestnuts, red and white guava, pomegranates, flaxseeds, dark chocolate and cocoa, coffee, tea, rose hip, olives, artichoke, dried herbs and beefsteak tongue mushrooms).
  Interventions: Other: Pomegranate Juice

INTERVENTIONS:
Other: Pomegranate Juice — Drinking 8 oz of pomegranate juice daily for 2 weeks.

SUMMARY:
Breast milk is universally recognized as the best food for newborns. Studies have scientifically shown that breastfeeding provides optimal nutrients for infants, strengthens their immune system, and improves mother-and-child bonding. Demonstrating health benefits of pomegranate consumption on infant health could lead to greater incentive for women to breast feed. The purpose of this research study is to determine whether pomegranate metabolites (products produced by breakdown) is secreted into breastmilk and whether they have an effect on breast-fed infants who are born vaginally.

DETAILED DESCRIPTION:
The study will require participants to continue with their usual diet and to avoid pomegranate juice (other than what is provided), berries (strawberries, blackberries, raspberries (red, black, yellow), cranberries), walnuts, pecans, hazelnuts, pecans, chestnuts, red and white guava, pomegranates, flaxseeds, dark chocolate and cocoa, coffee, tea, rose hip, olives, artichoke, dried herbs and beefsteak tongue mushrooms) . They will be asked to consume the pomegranate juice daily for 14 days. The pomegranate juice will be provided to participants. If the participants are unable to complete the study on the 14th day they will be asked to continue drinking the juice until they are able to complete the visit. For instance if day 14 falls on a Friday and they cannot come in until Monday participants will be asked to continue drinking the juice until Monday. Participants will be asked to collect 10ml (or 2 tsp) of breast milk; the collection materials will be provided, and participant will need to store the specimen in their home refrigerator and dropped off to the study site within 18-24 hours of the collection time. Participants will also be instructed to collect their stool and will be provided with the sterile collection materials and instructions for collection. Participants will be provided with a disposable cooler and ice packs to keep the specimen refrigerated during transport. Participants will also be provided with a urine collection container and asked to collect all of your urine over a 24-hour period (on 2 separate occasions). Lastly, infant stool and urine will also be collected using collection bags with an adhesive strip.

ELIGIBILITY:
Inclusion Criteria

* Postpartum 6 months with full term baby born vaginally and exclusively breast feeding
* In good health
* Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria

* No antibiotics or laxatives use during the 2 months before the study.
* Any subject consuming pre- or probiotics or anti-inflammatory medication
* Any subject with a screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
* Any subject who is unable or unwilling to comply with the study protocol.
* Allergic to pomegranate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Pomegranate Juice Metabolism | 2 weeks
  To examine the metabolism of pomegranate by analyzing blood, urine, breast milk and stool samples for ellagic acid and urolithin levels before and after administration of pomegranate extract for 2 weeks during breastfeeding in healthy mothers.
Microbiome | 2 weeks
  To determine whether pomegranate metabolites are bioavailable to breastfed infants by analyzing ellagic acid in urine and stool from infants of mothers consuming PJ.
Microbiome | 2 weeks
  To determine whether pomegranate metabolites are bioavailable to breastfed infants by analyzing urolithin in urine and stool from infants of mothers consuming PJ.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, Principal Investigator — UCLA Professor of Medicine
Locations (1):
- UCLA Center for Human Nutrition, 1000 Veteran Ave., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No